CLINICAL TRIAL: NCT02673515
Title: The Impact of Intermittent Fasting on Human Metabolism and Cell Autophagy
Acronym: InterFast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-2014-03
Record Dates: First submitted 2015-11-24; First posted 2016-02-04 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Excessive Diet Restriction
Keywords: Alternate Day Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alternate day fasting (Active Comparator): Subjects are requested to alternate fast for 4 weeks (alternate an ad libitum "feed day" with a 100% restriction "fast day").
  Interventions: Behavioral: Alternate day fasting
- control group (No Intervention): control group

INTERVENTIONS:
Behavioral: Alternate day fasting — Subjects are requested to fast every other day. Calorie free fluids are allowed.
  Arms: Alternate day fasting

SUMMARY:
InterFast is a Cohort study with an embedded randomized controlled pilot trial. Study participants will be healthy subjects and subjects who already practice Alternate Day Fasting. The trial will include 100 participants (50 Participants in Alternate Day Fasting group and 50 participants in the control group). Those participants in the control group will be asked to participate in a short randomized controlled trial, where they will be either allocated to an Alternative Day Fasting group or another control visit.

DETAILED DESCRIPTION:
Intermittent fasting is a dietary regimen defined by alternating fasting and "feeding" cycles. In addition to caloric restriction (a dietary regimen limited to a daily food intake lower than one's daily caloric needs) only, intermittent fasting seems to activate cell autophagy (cellular "recycling" program) which potentially increases cellular stress resistance and removes accumulated molecules that are potentially toxic. In fact, mice maintained on intermittent fasting without decreased overall food intake show effects on body weight reduction that equal and in some cases even exceed those of calorie restriction. However, additionally, intermittent fasting combined with even a high-fat diet in the feeding periods protects mice from obesity, hyperinsulinemia, hepatic steatosis, and inﬂammation compared to controls that are fed an ad libitum high-fat diet despite the same calorie intake, making this intermittent fasting regimen a promising approach to reduce morbidity and mortality in various species.

The best described and most widely practiced version of intermittent fasting is the "alternate day diet" or "alternate day fasting" (ADF). In animal models, ADF consists of an ad libitum "feed day" alternated with a 100% restriction "fast day". However in humans, this is often modified to allow a small amount of food consumption on the "fast day" (e.g. 25% of the individual´s energy needs). Findings from recent modified ADF studies showed significant reductions in body weight.

However, knowledge about the molecular effects of the alternate day diet on human metabolism or autophagy is still scarce since detailed analyses of molecular and metabolic parameters remain unexplored, especially in healthy individuals. The overarching aim of this research project is to elucidate in which extent alternate day fasting (and thereby intermittent fasting) influences human physiology in healthy individuals in both short and long term. The secondary objective of this study is to define novel molecular markers of aging and age-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index in the range of 22.0 - 27.0 kg/m2,
* Fasting blood glucose <110mg/dL (without medication)
* LDL-cholesterol <180 mg/dL (without medication)
* Blood pressure <140/90 mmHg (without medication)
* Stable weight (change <± 10%) for 3 months immediately prior to the study,
* No history of metabolic disorders or cardiovascular disease
* No acute or chronic inflammatory disorder
* No current medications to regulate blood sugar, blood pressure or lipids or hormones
* No heavy drinking (more than 15 drinks/week)
* No use of tobacco or recreational drugs within past 5 years
* No dietary restrictions (e.g. vegetarianism and vegan)

Exclusion Criteria:

* Known Malignancy
* Women who are pregnant, breast-feeding or trying to become pregnant
* History of any chronic disease process that could interfere with interpretation of study results
* Women or men on hormonal supplementation or anti-conceptive hormonal medication for at least 2 months
* Therapy with antidepressants within past 6 months
* Regular therapy with acetylsalicylic acid

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Medical University of Graz, Auenbruggerplatz 15; Frank Madeo, PhD, Study Chair — Karl Franzens University Graz, Austria; Thomas R Pieber, MD, Study Chair — Medical University Graz, Austria
Locations (1):
- Dept. of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tripolt NJ, Stekovic S, Aberer F, Url J, Pferschy PN, Schroder S, Verheyen N, Schmidt A, Kolesnik E, Narath SH, Riedl R, Obermayer-Pietsch B, Pieber TR, Madeo F, Sourij H. Intermittent Fasting (Alternate Day Fasting) in Healthy, Non-obese Adults: Protocol for a Cohort Trial with an Embedded Randomized Controlled Pilot Trial. Adv Ther. 2018 Aug;35(8):1265-1283. doi: 10.1007/s12325-018-0746-5. Epub 2018 Jul 25. PMID 30046988
- [Result] Stekovic S, Hofer SJ, Tripolt N, Aon MA, Royer P, Pein L, Stadler JT, Pendl T, Prietl B, Url J, Schroeder S, Tadic J, Eisenberg T, Magnes C, Stumpe M, Zuegner E, Bordag N, Riedl R, Schmidt A, Kolesnik E, Verheyen N, Springer A, Madl T, Sinner F, de Cabo R, Kroemer G, Obermayer-Pietsch B, Dengjel J, Sourij H, Pieber TR, Madeo F. Alternate Day Fasting Improves Physiological and Molecular Markers of Aging in Healthy, Non-obese Humans. Cell Metab. 2019 Sep 3;30(3):462-476.e6. doi: 10.1016/j.cmet.2019.07.016. Epub 2019 Aug 27. PMID 31471173
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After interviewing 462 adults for study eligibility based on previously set inclusion and exclusion criteria we have selected 60 representative study participants for the randomized controlled trial.
Groups:
- Control Group: participants in the control group should be remaining on their usual diet
Period: Overall Study
Arm/Group | Alternate Day Fasting | Control Group
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Lack of motivation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Day Fasting | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [42.5 to 55.0] | 50.5 [44.5 to 56.75] | 49 [43.25 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: per protocol analysis
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    Female | 17 | 17 | 34
    Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: per protocol analysis
  Participants
    number analyzed (Participants) | 28 | 29 | 57
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 28 | 29 | 57
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kg] — Population: per protocol analysis
  kg
    number analyzed (Participants) | 28 | 29 | 57
    (all) | 77.21 (10.25) | 75.93 (12.50) | 77.03 (11.90)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity (HOMA-IR)
Description: HOMA-Index was calculated by using the following formula:
  HOMA-IR= FPG(mmol/l)*FSI (U/l)/22.5 FSI=fasting serum insulin FPG=fasting plasma glucose
Time Frame: 4 weeks (from Baseline to 4 weeks)
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: no unit
Groups:
- Control Group: participants of the control group should be remaining on their usual diet
Arm/Group | Alternate Day Fasting | Control Group
Number analyzed (Participants) | 28 | 29
no unit | 0.05 (0.95) | 0.06 (0.80)

2. Primary Outcome: Insulin Sensitivity (QUICKI)
Description: QUICKI was calculated by using the following formula: QUICKI= log(FSI)+log (FPG) FSI=fasting serum insulin FPG=fasting plasma glucose
Time Frame: 4 weeks (from Baseline to 4 weeks)
Population: per protocol analysis
Measure: Median (Inter-Quartile Range); unit: no unit
Arm/Group | Alternate Day Fasting | Control Group
Number analyzed (Participants) | 28 | 29
no unit | 0 [-0.02 to 0.02] | 0 [-0.03 to 0.01]

3. Primary Outcome: Insulin Sensitivity (ISI-Index)
Description: ISI was calculated by using the following formula: ISI=0,222-0,00333 x BMI-0,0000779 x Ins120-0,000422 x age FSI=fasting serum insulin FPG=fasting plasma glucose
Time Frame: 4 weeks (from Baseline to 4 weeks)
Population: per protocol analysis
Measure: Median (Inter-Quartile Range); unit: no unit
Arm/Group | Alternate Day Fasting | Control Group
Number analyzed (Participants) | 28 | 29
no unit | 0 [0 to 0.01] | 0 [0.0 to 0.01]

4. Primary Outcome: Insulin Sensitivity (Matsuda-Index)
Description: Matsuda index was calculated by using the following formula:
  Matsuda-Index = 10000√(FPG∗FSI)∗(mean glucose*mean insulin) FSI=fasting serum insulin FPG=fasting plasma glucose
Time Frame: 4 weeks (from Baseline to 4 weeks)
Population: per protocol analysis
Measure: Median (Inter-Quartile Range); unit: no unit
Arm/Group | Alternate Day Fasting | Control Group
Number analyzed (Participants) | 28 | 29
no unit | -0.4 [-4.6 to 3.3] | -0.7 [-5.4 to 1.8]
Statistical Analysis 1: Comparison: Alternate Day Fasting vs Control Group; Comparison of changes from baseline to 4 weeks between groups was tested with student´s t-test or Mann Whitney-U-Test; Test type: Other; p = 0.797, t-test, 2 sided

5. Secondary Outcome: Blood Pressure (Systolic and Diastolic)
Description: Change of blood pressure from Baseline to 4 weeks
Time Frame: 4 weeks
Population: per protocol analysis
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Alternate Day Fasting | Control Group
Number analyzed (Participants) | 28 | 29
mmHg
  Systolic blood pressure | -4.5 [-7.75 to -0.5] | -1 [-6 to 7]
  Diastolic blood pressure | -2.5 [-4 to 1] | 0 [-3.5 to 2.5]

ADVERSE EVENTS:
Time Frame: During each study visit participants were asked about adverse events since the previous study visit. Adverse events were collected for 4 weeks (from study start to the end of the study).
Groups:
- Control Group: Participants in the control group should be remaining their normal diet
Arm/Group | Alternate Day Fasting | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02673515/Prot_000.pdf